CLINICAL TRIAL: NCT01387672
Title: Nitrates and Bone Turnover (NABT): Trial to Select the Best Nitrate Preparation
Brief Title: Nitrates and Bone Turnover; Nitrates and Bone Turnover Bisphosphonate Sub-Study
Acronym: NABT;NABT-B
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Toronto (Other)
Collaborators: The Physicians' Services Incorporated Foundation (Other); California Pacific Medical Center (Other); Sunnybrook Health Sciences Centre (Other); Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Sophie Jamal, Associate Professor/Endocrinologist, University of Toronto
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 062011
Record Dates: First submitted 2011-06-30; First posted 2011-07-04 (Estimated); Results first posted 2015-05-08 (Estimated); Last update posted 2015-05-08 (Estimated); Status verified 2015-05

CONDITIONS: Osteoporosis
Keywords: postmenopausal; osteoporosis; bone turnover; nitrate; headache
MeSH Terms: conditions — Osteoporosis; Headache | interventions — Nitrates

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- Nitrol (Active Comparator): Nitroglycerin Ointment 2% USP
  Interventions: Drug: Nitrates (NABT Main trial)
- Nitro-Dur (Active Comparator): Nitroglycerin Extended Release Patch 160mg
  Interventions: Drug: Nitrates (NABT Main trial)
- Nitrostat 1 (Active Comparator): Nitroglycerin 0.3mg Sublingual Tablet
  Interventions: Drug: Nitrates (NABT Main trial)
- Nitrostat 2 (Active Comparator): Nitroglycerin 0.6mg Sublingual Tablet
  Interventions: Drug: Nitrates (NABT Main trial)
- ISMO (Active Comparator): Isosorbide Mononitrate 20mg Oral Tablet
  Interventions: Drug: Nitrates (NABT Main trial)
- Placebo (Placebo Comparator): Placebo Ointment
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Nitrates (NABT Main trial) — nitroglycerin; isosorbide mononitrate
  Other Names: NABT-B Sub-Study: Nitroglycerin Ointment 2%: 15mg of NTG ointment for a 3 month period
  Arms: ISMO; Nitro-Dur; Nitrol; Nitrostat 1; Nitrostat 2
Other: Placebo — Placebo ointment
  Arms: Placebo

SUMMARY:
Purpose: NABT: To compare five widely available nitrate formulations: (1) 15 of nitroglycerin (NTG) ointment, (2) 0.3 mg and (3) 0.6 mg of sublingual NTG, (4) 20 mg of isosorbide mononitrate (an oral tablet), and (5) 160 mg of glycerol trinitrate (a patch), for their efficacy on markers of bone formation and resorption and for the incidence and severity of headache they cause.

Hypothesis: There is one ideal nitrate preparation which balances the clinical efficacy in bone remodeling against the common side effect of headache.

NABT-B: To determine if nitrates affect markers of bone formation (serum BALP and P1NP) and resorption (serum CTX and urine NTX) in women who have recently discontinued treatment with alendronate, risedronate or zoledronate.

ELIGIBILITY:
Inclusion Criteria:

NABT:

* Women aged 50 years and older whose last menstrual period occurred at least 3 years ago
* Women without a uterus will be eligible after age 55

NABT-B:

* Women aged 50 years and older whose last menstrual period occurred at least 3 years ago
* Women without a uterus will be eligible after age 55
* Previously treated with alendronate but stopped within 2 years of study commencement; or previously treated with risedronate but stopped within 1 year of study commencement; or previously treated with zoledronate.

Exclusion Criteria:

NABT:

* A previous fracture of the hip, wrist, spine or ankle within the last 3 months; or a diagnosis of osteoporosis;
* A history of bone disorders such as hyperparathyroidism or Paget's disease;
* Treatment within 12 months of study entry with any agent that may influence bone metabolism including any hormone, anti-estrogen or raloxifene and prednisone (equivalent to 5 mg/d for 12 months or greater);
* Treatment with any antiresorptive agent, including alendronate, risedronate, etidronate or denosumab use for at least four weeks within the last three years;
* Previous treatment with intravenous zoledronate or parathyroid hormone;
* Current treatment with nitrates;
* A history of migraine headaches;
* A history of angina or cardiovascular disease;
* Inability to give informed consent;
* Hypersensitivity to nitroglycerin.

NABT-B:

* A previous fracture of the hip, wrist, spine or ankle; or a self-reported diagnosis of osteoporosis;
* A history of bone disorders such as hyperparathyroidism or Paget's disease;
* Treatment within 12 months of study entry with any agent that may influence bone metabolism including any hormone, anti-estrogen or raloxifene and prednisone (equivalent to 5 mg/d for 12 months or greater);
* Treatment with etidronate or denosumab use for at least four weeks within the last three years and any previous treatment with parathyroid hormone;
* Current treatment with nitrates;
* A history of migraine headaches;
* A history of angina or cardiovascular disease;
* Inability to give informed consent;
* Hypersensitivity to nitroglycerin.

Min Age: 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 265 (Actual)
Dates: Start 2011-09; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sophie A Jamal, MD,PhD,FRCPC, Principal Investigator — Women's College Research Institute/Women's College Hospital
Locations (1):
- Women's College Research Institute/Women's College Hospital, Toronto, Ontario, Canada

REFERENCES:
- [Background] Jamal SA, Hamilton CJ, Eastell R, Cummings SR. Effect of nitroglycerin ointment on bone density and strength in postmenopausal women: a randomized trial. JAMA. 2011 Feb 23;305(8):800-7. doi: 10.1001/jama.2011.176. PMID 21343579 (Retraction: PMID 26719994 Eastell R, Hamilton CJ, Cummings SR. JAMA. 2016 Jan 26;315(4):418-9)
- [Background] Jamal SA, Goltzman D, Hanley DA, Papaioannou A, Prior JC, Josse RG. Nitrate use and changes in bone mineral density: the Canadian Multicentre Osteoporosis Study. Osteoporos Int. 2009 May;20(5):737-44. doi: 10.1007/s00198-008-0727-7. Epub 2008 Sep 18. PMID 18800179 (Retraction: PMID 27909783 Osteoporos Int. 2016 Dec 1;:)
- [Background] Jamal SA, Cummings SR, Hawker GA. Isosorbide mononitrate increases bone formation and decreases bone resorption in postmenopausal women: a randomized trial. J Bone Miner Res. 2004 Sep;19(9):1512-7. doi: 10.1359/JBMR.040716. Epub 2004 Jul 26. PMID 15312252
- [Background] Jamal SA, Browner WS, Bauer DC, Cummings SR. Intermittent use of nitrates increases bone mineral density: the study of osteoporotic fractures. J Bone Miner Res. 1998 Nov;13(11):1755-9. doi: 10.1359/jbmr.1998.13.11.1755. PMID 9797485
- [Background] Wimalawansa SJ, Grimes JP, Wilson AC, Hoover DR. Transdermal nitroglycerin therapy may not prevent early postmenopausal bone loss. J Clin Endocrinol Metab. 2009 Sep;94(9):3356-64. doi: 10.1210/jc.2008-2225. Epub 2009 Jun 23. PMID 19549739
- [Derived] Bucur RC, Reid LS, Hamilton CJ, Cummings SR, Jamal SA. Nitrates and bone turnover (NABT) - trial to select the best nitrate preparation: study protocol for a randomized controlled trial. Trials. 2013 Sep 8;14:284. doi: 10.1186/1745-6215-14-284. PMID 24010992

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Initial run-in period-subjects received, in random order, each of the 5 nitrate formulations for 2 days with a 2 day wash out period between formulations. There were 265 subjects enrolled in the run-in phase of the study. Out of those, 229 subjects entered the treatment phase of the study, where they were randomized to one of the 6 treatment arms.
Groups:
- ISMO - Treatment Arm 1: Isosorbide Mononitrate 20mg Oral Tablet
  Nitrates (NABT Main trial)
- Patch (Nitro-Dur) - Treatment Arm 2: Nitroglycerin Extended Release Patch 160mg
  Nitrates (NABT Main trial)
- Ointment (Nitrol) - Treatment Arm 3: Nitroglycerin Ointment 2% USP
  Nitrates (NABT Main trial)
- 0.3 Sublingual (Nitrostat 1) - Treatment Arm 4: Nitroglycerin 0.3mg Sublingual Tablet
  Nitrates (NABT Main trial)
- 0.6 Sublingual (Nitrostat 2) - Treatment Arm 5: Nitroglycerin 0.6mg Sublingual Tablet
  Nitrates (NABT Main trial)
- Placebo Ointment - Treatment Arm 6: Placebo Ointment
  Nitrates (NABT Main trial)
Period: Overall Study
Arm/Group | ISMO - Treatment Arm 1 | Patch (Nitro-Dur) - Treatment Arm 2 | Ointment (Nitrol) - Treatment Arm 3 | 0.3 Sublingual (Nitrostat 1) - Treatment Arm 4 | 0.6 Sublingual (Nitrostat 2) - Treatment Arm 5 | Placebo Ointment - Treatment Arm 6
Started | 39 | 38 | 38 | 39 | 38 | 37
Completed | 32 | 31 | 33 | 35 | 34 | 37
Not Completed | 7 | 7 | 5 | 4 | 4 | 0

BASELINE CHARACTERISTICS:
Groups:
- Placebo Ointment - Treatment Arm 6: Placebo Ointment
  Placebo: Placebo ointment Nitrates (NABT Main trial)
- Total: Total of all reporting groups
Arm/Group | ISMO - Treatment Arm 1 | Patch (Nitro-Dur) - Treatment Arm 2 | Ointment (Nitrol) - Treatment Arm 3 | 0.3 Sublingual (Nitrostat 1) - Treatment Arm 4 | 0.6 Sublingual (Nitrostat 2) - Treatment Arm 5 | Placebo Ointment - Treatment Arm 6 | Total
Number analyzed (Participants) | 39 | 38 | 38 | 39 | 38 | 37 | 229
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 19 | 21 | 20 | 23 | 23 | 20 | 126
  >=65 years | 20 | 17 | 18 | 16 | 15 | 17 | 103
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39 | 38 | 38 | 39 | 38 | 37 | 229
  Male | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Canada | 39 | 38 | 38 | 39 | 38 | 37 | 229

OUTCOME MEASURES:

1. Primary Outcome: Bone Turnover Markers
Description: Markers of Bone Formation:
  * Serum Procollagen type 1 amino- terminal propeptide (P1NP)
  * Serum Osteocalcin (OC)
  * Serum Bone-specific alkaline phosphatase (BALP)
  Markers of Bone Resorption:
  - Serum C-telopeptides of collagen cross-links (CTX)
Time Frame: 3 months
Population: One subject from the Treatment Arm 3 had outlier bone turnover markers values and was excluded from the analysis. Total number of subjects analyzed in Treatment Arm 3 was therefore 32.
Measure: Mean (Standard Deviation); unit: Percent change from baseline
Arm/Group | ISMO - Treatment Arm 1 | Patch (Nitro-Dur) - Treatment Arm 2 | Ointment (Nitrol) - Treatment Arm 3 | 0.3 Sublingual (Nitrostat 1) - Treatment Arm 4 | 0.6 Sublingual (Nitrostat 2) - Treatment Arm 5 | Placebo Ointment - Treatment Arm 6
Number analyzed (Participants) | 32 | 31 | 32 | 35 | 34 | 37
Percent change from baseline
  P1NP | -4.627 (16.191) | -0.405 (20.289) | -4.297 (16.236) | -6.126 (16.093) | 2.941 (36.843) | -1.635 (16.749)
  OC | -3.244 (12.049) | 3.796 (33.601) | -4.481 (14.823) | 1.046 (21.818) | 1.033 (17.931) | 4.247 (22.088)
  BALP | -5.023 (11.824) | -0.541 (20.738) | -7.426 (11.056) | -7.000 (19.011) | -3.686 (17.435) | -1.648 (21.523)
  CTX | -5.844 (26.084) | -1.025 (32.163) | -9.699 (27.299) | -0.666 (37.945) | -1.380 (52.248) | -1.783 (28.063)

2. Secondary Outcome: Headache
Description: Severity of headaches. Subjects recorded the severity of headaches upon awakening every day during the run-in phase using a visual analogue scale (VAS). The scale is represented by a line (continuum) 10 cm long. Subjects were asked to make a vertical line along the continuum to indicate the severity of their headache each morning upon awakening. The score is recorded in cm from "0" to "10". A vertical line marked at "0" means no headache (score recorded = "0"), a vertical line marked at "10" means a terrible headache (score recorded = "10").
Time Frame: Run-in phase - 2 days
Population: The mean headache score considering all subjects in each of the treatment/formulation group was calculated.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Run-in Phase: During the run-in phase subjects received, in random order, each of the 5 nitrate formulations for 2 days with a 2 day wash out period between formulations. The severity of headaches was recorded, by subjects, upon awakening, every day during the run in phase using a visual analog scale (VAS).
Arm/Group | Run-in Phase
Number analyzed (Participants) | 238
score on a scale
  ISMO | 2.1 (2.64)
  Patch | 3.1 (2.98)
  Ointment | 1.5 (2.12)
  0.3 Sublingual | 0.36 (1.18)
  0.6 Sublingual | 0.6 (1.62)

ADVERSE EVENTS:
Time Frame: The Adverse Events are reported for the 3 months treatment phase of the study, once the patients were randomized to a specific treatment arm (ISMO - Arm 1; Patch - Arm 2; Ointment - Arm 3; 0.3 Sublingual - Arm 4; 0.6 Sublingual - Arm 5 or Placebo - Arm 6)
Groups:
- Placebo Ointment- Treatment Arm 6: Placebo Ointment
  Placebo: Placebo ointment Nitrates (NABT Main trial)
Arm/Group | ISMO - Treatment Arm 1 | Patch (Nitro-Dur) - Treatment Arm 2 | Ointment (Nitrol) - Treatment Arm 3 | 0.3 Sublingual (Nitrostat 1) - Treatment Arm 4 | 0.6 Sublingual (Nitrostat 2) - Treatment Arm 5 | Placebo Ointment- Treatment Arm 6
Serious Adverse Events (participants affected / at risk) | 0/39 | 0/38 | 0/38 | 1/39 | 1/38 | 0/37
Other Adverse Events (participants affected / at risk) | 17/39 | 21/38 | 17/38 | 10/39 | 12/38 | 6/37
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ISMO - Treatment Arm 1 (N=39) | Patch (Nitro-Dur) - Treatment Arm 2 (N=38) | Ointment (Nitrol) - Treatment Arm 3 (N=38) | 0.3 Sublingual (Nitrostat 1) - Treatment Arm 4 (N=39) | 0.6 Sublingual (Nitrostat 2) - Treatment Arm 5 (N=38) | Placebo Ointment- Treatment Arm 6 (N=37)
Transient Global Amnesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Stroke (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ISMO - Treatment Arm 1 (N=39) | Patch (Nitro-Dur) - Treatment Arm 2 (N=38) | Ointment (Nitrol) - Treatment Arm 3 (N=38) | 0.3 Sublingual (Nitrostat 1) - Treatment Arm 4 (N=39) | 0.6 Sublingual (Nitrostat 2) - Treatment Arm 5 (N=38) | Placebo Ointment- Treatment Arm 6 (N=37)
Headache (Nervous system disorders) | 17 (17) | 21 (21) | 17 (17) | 10 (10) | 12 (112) | 6 (6)
Dizziness (Nervous system disorders) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0) | 2 (2) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No